CLINICAL TRIAL: NCT01095055
Title: A Phase I Study to Assess the Safety and Immunogenicity of New Malaria Vaccine Candidates AdCh63 AMA1 Alone and With MVA AMA1
Brief Title: A Study of AdCh63 AMA1 Alone and With MVA AMA1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Prof Adrian Hill, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC036
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): AdCh63 AMA1
  Interventions: Biological: AdCh63 AMA1
- Group 2 (Experimental): AdCh63 AMA1 followed by MVA AMA1
  Interventions: Biological: AdCh63 AMa1 and MVA AMA1

INTERVENTIONS:
Biological: AdCh63 AMA1 — Group 1A - single dose of AdCH63 AMA1 5x10^9 vp intramuscularly Group 2A - single dose of AdCH63 AMA1 5x10^10 vp intramuscularly
  Other Names: Simian adenovirus expressing malaria antigen AMA1
  Arms: Group 1
Biological: AdCh63 AMa1 and MVA AMA1 — Group 1B - single dose of AdCH63 AMA1 5x10^9 vp intramuscularly and single dose of MVA AMA1 5x10^8 pfu 8 weeks later intramuscularly Group 2B - single dose of AdCH63 AMA1 5x10^10 vp intramuscularly and single dose of MVA AMA1 5x10^8 pfu 8 weeks later intramuscularly
  Other Names: Simian adenovirus, modified vaccinia Ankara virus expressing malaria antigen AMA1
  Arms: Group 2

SUMMARY:
This is an open label phase I study, to assess the safety of a novel malaria vaccine, AdCh63 AMA1, simian adenovirus encoding Plasmodium falciparum blood stage antigen, Apical Membrane Antigen -1. All volunteers recruited will be healthy adults. They will be primed with various doses of AdCh63 AMA1 administered intramuscularly. Some of the volunteers will receive a booster vaccination with MVA AMA1 administered via intramuscular route. Safety data will be collected for each of the eight regimens. Secondary aims of this study will be to assess the immune responses generated by each of these regimes.

DETAILED DESCRIPTION:
AMA1 is a type I integral membrane protein. It is produced by mature P. falciparum schizonts in infected erythrocytes AMA1 has become a leading candidate vaccine antigen. This is based on several facts, most notably that in several field studies an association was found between antibodies to the ectodomain of AMA1 and protection against clinical malaria. Also, in the Gambia, presence of antibodies to AMA1 and MSP-1 has been shown to enhance clearance of chloroquine resistant parasites in vivo.

There are a number of trials currently ongoing in Oxford which are aimed at examining a simian adenovirus as a delivery vehicle and liver and blood stage malaria antigens as inserts. AdCh63 is currently in use with the MSP-1 insert, a blood stage antigen, in a phase I dose escalation clinical trial in Oxford (VAC037 / GTAC 166). The trial design includes AdCh63 MSP-1 administered alone and with MVA MSP-1 as part of a heterologous prime boost schedule, with sporozoite challenge of 3 volunteers in the higher dose group. At the most recent interim analysis, AdCh63 MSP-1 demonstrates an excellent safety profile.

Also, AdCh63 is currently in use with the ME-TRAP insert, a liver stage antigen in a phase I dose escalation clinical trial in Oxford, (VAC033 / GTAC133) and a phase I/IIa trial with sporozoite challenge (MAL034 / OXREC: 09/H064/9). AdCh63 ME-TRAP has been administered alone and with MVA ME-TRAP as part of a heterologous prime boost schedule at various doses with excellent safety and immunogenicity to 87 volunteers at time of interim analysis.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults aged 18 to 50 years

* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective barrier contraception during the study and a negative pregnancy test on the day(s) of vaccination
* For males only to use barrier contraception until three months after the last vaccination
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period

* Prior receipt of a recombinant adenoviral vaccine.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products, Kathon.
* History of clinically significant contact dermatitis
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study.
* Any history of malaria or
* Travel to a malaria endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety of AdCh63 administered alone, and combinedwith MVA AMA1 | Up to 6 months following the last vaccination
  To assess the safety in healthy volunteers of two candidate malaria vaccines, AdCh63 AMA1 with MVA AMA1 in a prime-boost regimen. The safety of AdCh63 administered alone, and combined with MVA AMA1 will be assessed. The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events.

SECONDARY OUTCOMES:
The level of immune response induced by vaccination with AdCh63 AMA1, when administered as a single vaccination and sequentially with MVA AMA1 | Up to 6 moths following the last vaccination
  To assess the level of immune response induced by vaccination with AdCh63 AMA1, when administered as a single vaccination and sequentially with MVA AMA1

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, Principal Investigator — Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Churchill Hospital
Locations (2):
- United Kingdom (2):
  - Hospital for Tropical Diseases, London
  - Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Old Road, Headington, Oxford

REFERENCES:
- [Derived] Sheehy SH, Duncan CJ, Elias SC, Biswas S, Collins KA, O'Hara GA, Halstead FD, Ewer KJ, Mahungu T, Spencer AJ, Miura K, Poulton ID, Dicks MD, Edwards NJ, Berrie E, Moyle S, Colloca S, Cortese R, Gantlett K, Long CA, Lawrie AM, Gilbert SC, Doherty T, Nicosia A, Hill AV, Draper SJ. Phase Ia clinical evaluation of the safety and immunogenicity of the Plasmodium falciparum blood-stage antigen AMA1 in ChAd63 and MVA vaccine vectors. PLoS One. 2012;7(2):e31208. doi: 10.1371/journal.pone.0031208. Epub 2012 Feb 21. PMID 22363582